CLINICAL TRIAL: NCT06064032
Title: Comparing The Effects Of Cognitive Behavioral Therapy And Motor Learning Technique in Adults With Attention Deficit Hyperactivity Disorder.
Brief Title: Cognitive Behavioral Therapy And Motor Learning Technique Among Attention Deficit Hyperactivity Disorder Adults
Acronym: ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSAHS 2023/03
Record Dates: First submitted 2023-09-08; First posted 2023-10-03 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The subjects in the experimental group will be given a 10 minute session of Progressive Muscle Relaxation (PMR), 2 minutes deep breathing exercises,3 minutes training for life style modification which includes the use of planners, setting alarms, breaking a difficult task into parts, positive reinforcement and communication combined with a 3 minute session of drawing a specific pattern with installing pegs on pegboard, 2 minutes session of balance board training, 3 min session of solving jigsaw puzzles, 1 minute session of squeezing a ball with maximum repetition and 1 minute session of finding beads in puttey. . After the completion of therapy, the participants will be assessed by the proforma used to diagnose the ADHD and their respective scores will be noted and compared with the previous ones.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All the recruited participants will be assigned serial numbers and will be randomly divided into two groups using lottery method.The participants file will be prepared and will be kept under custody of Principal Investigator. List will be provided to outcome assessor for respected treatment and directing the participant to care giver. Outcome assessor will collect the data before and after each session in a separate assigned space. Score will be recorder on 1st , 7th and 15th day of treatment session by the investigator. After that respected scores will be computed & analyzed by the outcome assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive behvioral therapy (Active Comparator): The subjects in the control group will be given a 10 minute session of Progressive Muscle Relaxation (PMR) 2 minutes deep breathing exercises and 3 minutes training for life style modification which includes the use of planners, setting alarms, breaking a difficult task into parts, positive reinforcement and communication. This would be taught for 15 days at one day interval.
  Interventions: Behavioral: cognitive behavioral therapy
- motor learning techniques (Experimental): The subjects in the experimental group will be given a 10 minute session of Progressive Muscle Relaxation (PMR), 2 minutes deep breathing exercises,3 minutes training for life style modification which includes the use of planners, setting alarms, breaking a difficult task into parts, positive reinforcement and communication combined with a 3 minute session of drawing a specific pattern with installing pegs on pegboard, 2 minutes session of balance board training, 3 min session of solving jigsaw puzzles, 1 minute session of squeezing a ball with maximum repetition and 1 minute session of finding beads in puttey.
  This would be taught for 15 days at one day interval.
  Interventions: Behavioral: cognitive behavioral therapy; Behavioral: Motor Learning Techniques

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — In control group there is 10 min session of PMR, 2 min deep breathing exercises,3 min training for life style modification which include use of planner, setting alarms breaking a task into parts positive reinforcement and communication.
Behavioral: Motor Learning Techniques — In experimental group, participants will be given a 10 min PMR ,2 min deep breathing exercises, 3 min training for life style modification which include the use of planners setting alarms, breaking a difficult task into parts, positive reinforcement and communication combined with 3 min session of drawing a specific pattern with installing pegs on pegboard, 2 min session of balance board training, 3 min session of jigsaw puzzle training, 1 min session of squeezing a ball with maximum repetition and 1 min session of finding beads in puttey.
  Arms: motor learning techniques

SUMMARY:
The aim of our study to compare the effect of cognitive behavioral therapy and motor learning techniques in adults with Attention Deficit Hyperactivity Disorder. and help the adults to address and revise cognitive distortions and habits affecting your productivity and emotional mindset.participant allocated to control group will be asked to perform cognitive behavioural therapy and participants allocated to experimental group will be asked to perform motor learning activities and cognitive behavioral therapy.

DETAILED DESCRIPTION:
Attention deficit disorder/hyperactivity (ADHD) among adults is a frequent but under-diagnosed clinical situation. Attention deficit hyperactivity disorder prevails from childhood to adulthood and most of the adults suffering from this disorder were the same who went through this syndrome in their childhood.

Basically, ADHD has 3 main types in adults: In attentive ADHD with lack of attention to task, Impulsive ADHD with lack of decision-making skills and Combination of type 1 and 2.

Risk factors that lead to this disorder include: genetics ,environmental factors and developmental factors.

Meyer and Sag olden also found motor impairments in all three subtypes but they reported the strongest motor control problems and difficulty with gross motor skills in the combined type of ADHD.

ADHD significantly impairs multiple aspects of life, leading to educational underachievement, unemployment, unsuccessful marriage and criminality, etc. Moreover, ADHD shows significant correlations with a wide range of co-morbid psychiatric disorders, including effective disorders, antisocial personality disorder, self-harm, substance misuse, placing a considerable burden on society and family .

This syndrome include difficulty in performing activities of daily living, difficulty in making decisions and loss of attention while performing a task. They feel trouble in following and remembering plans, important events and daily tasks.

Men and women suffering from ADHD also encounter some motor control problems in their lives like lack of dexterity, gripping and fine motor skills.

A random affect meta-analysis of these studies showed that the global prevalence of ADHD in children and adolescents was 8.0 %.

Attention deficit hyperactivity disorder (ADHD) is recognised as the most common neurodevelopmental disorder of childhood. A frequently cited study by Polanszky of 2007 reported a worldwide ADHD prevalence estimate of 5.3%.

The overall Canadian ADHD prevalence estimate is similar to worldwide estimates for adults that is 5.3%. Estimates for children include 7.5% in Australia and 10.2% in the United States.

Two studies on adolescents in Africa provided estimates of 7.5%. A 2021 survey conducted in the United States, for example, found an ADHD prevalence rate for adults of 4.25% One German study on children and adolescents combined provides an estimate of 6.1.

In china there is 7.5% of rural students are at risk of ADHD. A study at India showed that 24.3% of the total study population had the presence of adult ADHD.

In Pakistan, a study conducted on 1889 patients showed almost 11% patients had diagnosis of ADHD after a screening questionnaire from their consultant.

After analyzing the properties of the ASRS (sensitivity: 83.3% specificity: 66.1%), we administered the Adult ADHD Self-Report Scale (ASRS) to detect the participants with attention deficit hyperactive disorder.

To assess the cognitive part of ADHD we use MOCA test also known as Montreal cognitive assessment which involves a picture-based marking system.

Perceptual-motor training is the best physical activity intervention for children with ADHD regarding motor ability and working memory. This type of training combines physical activities such as coordination, balance, and strength with perceptual tasks.

Longer exercise intervention (motor learning techniques) duration was consistently associated with larger effect sizes (g .627). Results suggest that exercise has a modest positive impact on ADHD functional outcomes, such as executive functions and motor skills, with longer interventions yielding better results.

Cognitive behavioral therapy can be given individually as well as in groups to treat main behavioral and cognitive impairments in patients of different age groups and more importantly with attention deficit hyperactivity disorder.

A systematic review showed that CBT was superior to control and superior to active control groups with a small to moderate effect size (SMD 0.43, 95% CI [0.14, 0.71], p .004).

CBT reduced ADHD symptoms (self and independently rated) compared with the control treatment(s).

Cognitive-motor training is an intervention that integrates cognitive and motor tasks to promote an individual's physical and mental health. It has been shown that performing two or more cognitive-motor tasks simultaneously, such as computation in postural training and movement under computer games, will contribute more to improvements in cognitive domains compared to single-task training.

Attention-deficit hyperactivity disorder also known as ADHD, is a neurobiological disorder that affects children and adults. It is associated with increased activity level and lack of attention regarding daily activities of living.

Cognitive behavioural therapy is method to encounter the negative thoughts and converting them into positive ones by using the method of reinforcement. Also, it can help people change the way they think about their problems.

Motor learning strategies can be applied in such people. Motor learning techniques are used to enhance someone's ability to perform a task more effectively and efficiently. They progress from a stage of dependency to automacity. These techniques are used for the acquisition and modification of a task to make it more effective.

ELIGIBILITY:
Inclusion Criteria:

* Medical & Allied health students, both male and females, aged between (18-29).
* Students who will score less than 26 out of 30 in MOCA test

Exclusion Criteria:

•Students with any history of systemic disease.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparing the Effect of Cognitive Behavioral Therapy and Motor Learning Techniques in Adults with Attention Deficit Hyperactivity Disorder. | 1-Month
  After analyzing the properties of the Adult self report scale( sensitivity: 83.3%, specificity:66.1 %) we administered adult self report scale to detect the participants with attention deficit hyperactivity disorder. In this 0 will be considered as the normal score( 14 or 14 above will be considered positive for attention deficit hyperactivity disorder) and 72 shows the severity of attention deficit hyperactivity disorder participants.

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Abbas, DPT, Principal Investigator — Shalamar Medical and Dental College; Meesha Naseer, DPT, Principal Investigator — Shalamar Medical and Dental College

REFERENCES:
- [Background] Weibel S, Menard O, Ionita A, Boumendjel M, Cabelguen C, Kraemer C, Micoulaud-Franchi JA, Bioulac S, Perroud N, Sauvaget A, Carton L, Gachet M, Lopez R. Practical considerations for the evaluation and management of Attention Deficit Hyperactivity Disorder (ADHD) in adults. Encephale. 2020 Feb;46(1):30-40. doi: 10.1016/j.encep.2019.06.005. Epub 2019 Oct 11. PMID 31610922
- [Background] Salvi V, Migliarese G, Venturi V, Rossi F, Torriero S, Vigano V, Cerveri G, Mencacci C. ADHD in adults: clinical subtypes and associated characteristics. Riv Psichiatr. 2019 Mar-Apr;54(2):84-89. doi: 10.1708/3142.31249. PMID 30985833
- [Background] Palladino VS, McNeill R, Reif A, Kittel-Schneider S. Genetic risk factors and gene-environment interactions in adult and childhood attention-deficit/hyperactivity disorder. Psychiatr Genet. 2019 Jun;29(3):63-78. doi: 10.1097/YPG.0000000000000220. PMID 30741787
- [Background] Lelong M, Zysset A, Nievergelt M, Luder R, Gotz U, Schulze C, Wieber F. How effective is fine motor training in children with ADHD? A scoping review. BMC Pediatr. 2021 Nov 4;21(1):490. doi: 10.1186/s12887-021-02916-5. PMID 34736439
- [Background] Song P, Zha M, Yang Q, Zhang Y, Li X, Rudan I; Global Health Epidemiology Reference Group (GHERG). The prevalence of adult attention-deficit hyperactivity disorder: A global systematic review and meta-analysis. J Glob Health. 2021 Feb 11;11:04009. doi: 10.7189/jogh.11.04009. PMID 33692893
- [Background] Thorell LB, Holst Y, Sjowall D. Quality of life in older adults with ADHD: links to ADHD symptom levels and executive functioning deficits. Nord J Psychiatry. 2019 Oct;73(7):409-416. doi: 10.1080/08039488.2019.1646804. Epub 2019 Aug 5. PMID 31380715
- [Background] Fietsam AC, Tucker JR, Kamath MS, Huang-Pollock C, Wang Z, Neely KA. Manual dexterity and strength and in young adults with and without Attention-Deficit/Hyperactivity Disorder (ADHD). Neurosci Lett. 2022 Jan 1;766:136349. doi: 10.1016/j.neulet.2021.136349. Epub 2021 Nov 14. PMID 34785312
- [Background] Ayano G, Demelash S, Gizachew Y, Tsegay L, Alati R. The global prevalence of attention deficit hyperactivity disorder in children and adolescents: An umbrella review of meta-analyses. J Affect Disord. 2023 Oct 15;339:860-866. doi: 10.1016/j.jad.2023.07.071. Epub 2023 Jul 24. PMID 37495084
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] Graetz BW, Sawyer MG, Hazell PL, Arney F, Baghurst P. Validity of DSM-IVADHD subtypes in a nationally representative sample of Australian children and adolescents. J Am Acad Child Adolesc Psychiatry. 2001 Dec;40(12):1410-7. doi: 10.1097/00004583-200112000-00011. PMID 11765286
- [Background] Ayano G, Yohannes K, Abraha M. Epidemiology of attention-deficit/hyperactivity disorder (ADHD) in children and adolescents in Africa: a systematic review and meta-analysis. Ann Gen Psychiatry. 2020 Mar 13;19:21. doi: 10.1186/s12991-020-00271-w. eCollection 2020. PMID 32190100
- [Background] London AS, Landes SD. Cohort Change in the Prevalence of ADHD Among U.S. Adults: Evidence of a Gender-Specific Historical Period Effect. J Atten Disord. 2021 Apr;25(6):771-782. doi: 10.1177/1087054719855689. Epub 2019 Jun 13. PMID 31189421
- [Background] Pang X, Wang H, Dill SE, Boswell M, Pang X, Singh M, Rozelle S. Attention Deficit Hyperactivity Disorder (ADHD) among elementary students in rural China: Prevalence, correlates, and consequences. J Affect Disord. 2021 Oct 1;293:484-491. doi: 10.1016/j.jad.2021.06.014. Epub 2021 Jun 18. PMID 34280772
- [Background] Samal B, Senjam G, Ravan JR, Ningombam HS, Das RC, Das SK. Prevalence of adult ADHD in patients with substance use disorder in North East India. Ind Psychiatry J. 2022 Jul-Dec;31(2):214-220. doi: 10.4103/ipj.ipj_250_21. Epub 2022 Aug 18. PMID 36419685
- [Background] Khan S, Qayyum R, Iqbal J. Prevalence of Autism Spectrum Disorders (ASD) and Attention Deficit Hyperactivity Disorders (ADHD) among Adult Psych. Pakistan Armed Forces Medical Journal. 201969(2):419-23
- [Background] Roncero C, Ortega L, Perez-Pazos J, Lligona A, Abad AC, Gual A, Sorribes M, Grau-Lopez L, Casas M, Daigre C. Psychiatric Comorbidity in Treatment-Seeking Alcohol Dependence Patients With and Without ADHD. J Atten Disord. 2019 Oct;23(12):1497-1504. doi: 10.1177/1087054715598841. Epub 2015 Aug 12. PMID 26269096
- [Background] Moyano S, Berrios W, Gandino I, Soriano E, Rosa J. POS0025 PREVALENCE OF ATTENTION DEFICIT HYPERACTIVITY DISORDER AMONG ADULT PATIENTS WITH FIBROMYALGIA. BMJ Publishing Group Ltd 2022.
- [Background] Hattabi S, Bouallegue M, Ben Yahya H, Bouden A. Rehabilitation of ADHD children by sport intervention: a Tunisian experience. Tunis Med. 2019 Jul;97(7):874-881. PMID 31872398
- [Background] Vysniauske R, Verburgh L, Oosterlaan J, Molendijk ML. The Effects of Physical Exercise on Functional Outcomes in the Treatment of ADHD: A Meta-Analysis. J Atten Disord. 2020 Mar;24(5):644-654. doi: 10.1177/1087054715627489. Epub 2016 Feb 9. PMID 26861158
- [Background] Anastopoulos AD, Langberg JM, Eddy LD, Silvia PJ, Labban JD. A randomized controlled trial examining CBT for college students with ADHD. J Consult Clin Psychol. 2021 Jan;89(1):21-33. doi: 10.1037/ccp0000553. PMID 33507774
- [Background] Young Z, Moghaddam N, Tickle A. The Efficacy of Cognitive Behavioral Therapy for Adults With ADHD: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Atten Disord. 2020 Apr;24(6):875-888. doi: 10.1177/1087054716664413. Epub 2016 Aug 22. PMID 27554190
- [Background] Dittner AJ, Hodsoll J, Rimes KA, Russell AJ, Chalder T. Cognitive-behavioural therapy for adult attention-deficit hyperactivity disorder: a proof of concept randomised controlled trial. Acta Psychiatr Scand. 2018 Feb;137(2):125-137. doi: 10.1111/acps.12836. Epub 2017 Dec 27. PMID 29282731
- [Background] Amini A, Vaezmousavi M, Shirvani H. The effectiveness of cognitive-motor training on reconstructing cognitive health components in older male adults, recovered from the COVID-19. Neurol Sci. 2022 Feb;43(2):1395-1403. doi: 10.1007/s10072-021-05502-w. Epub 2021 Jul 30. PMID 34328579
- [Background] Luo Y, Weibman D, Halperin JM, Li X. A Review of Heterogeneity in Attention Deficit/Hyperactivity Disorder (ADHD). Front Hum Neurosci. 2019 Feb 11;13:42. doi: 10.3389/fnhum.2019.00042. eCollection 2019. PMID 30804772
- [Background] Pan MR, Huang F, Zhao MJ, Wang YF, Wang YF, Qian QJ. A comparison of efficacy between cognitive behavioral therapy (CBT) and CBT combined with medication in adults with attention-deficit/hyperactivity disorder (ADHD). Psychiatry Res. 2019 Sep;279:23-33. doi: 10.1016/j.psychres.2019.06.040. Epub 2019 Jun 29. PMID 31280035
- [Background] Xie Y, Gao X, Song Y, Zhu X, Chen M, Yang L, Ren Y. Effectiveness of Physical Activity Intervention on ADHD Symptoms: A Systematic Review and Meta-Analysis. Front Psychiatry. 2021 Oct 26;12:706625. doi: 10.3389/fpsyt.2021.706625. eCollection 2021. PMID 34764893